CLINICAL TRIAL: NCT03246646
Title: Telephone Coaching of Family Members of Veterans With Substance Abuse Problems
Acronym: VA-CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D2070-P
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Substance Abuse
Keywords: Substance Abuse; Alcohol Abuse
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: The intervention will be approximately 12, 30-45 min. telephone sessions, every 2-3 weeks, and will last 4-6 months. The Coach helps the participant individualize the content of a web-based course (VA-CRAFT) based on an intervention to encourage a loved one to seek treatment for substance abuse. The VA-CRAFT course has 8 modules that follow the original CRAFT intervention: 1) Introduction, 2) Overview, 3) Getting Started: Safety Planning, 4) Understanding substance abuse, 5) How to respond to substance abuse, 6) Rebuilding your life together, 7) Helping someone consider treatment, 8) Wrapping up. The goals include understanding triggers and long-term reinforcement of substance misuse, ignoring unhealthy behaviors and rewarding healthy behaviors, getting support, and how to help the CSO caller help the Veteran enter treatment. The participants in the active intervention will be compared to a treatment as usual, matched comparator group drawn from regular clinical operations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coaching + VA CRAFT (Experimental): Telephone coaching along with web-based CRAFT course
  Interventions: Behavioral: Coaching
- Treatment as usual (Other): Treatment as usual matched comparison
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Telephone coaching was provided in a series of telephone based sessions with CSO participants

SUMMARY:
This project will develop and pilot test an enhanced, telephone "coaching" intervention to help family members concerned about a Veteran of the wars in Iraq or Afghanistan who needs to seek treatment for a substance abuse problem.

DETAILED DESCRIPTION:
The investigators will first develop a detailed manual for Coaching-CRAFT, which will be a telephone-based model of coaching that uses the web-version of an intervention already developed and available to the investigators. The investigators will conduct a preliminary nonrandomized feasibility trial of the use of Coaching-CRAFT with a sample of 50 family member callers recruited from VA's Coaching Into Care call center. Later in the study, the investigators will recruit up to 50 Veterans whose family members also participated in this study. Since the 'Coaching Into Care' telephone-based call center located at the Corporal Michael J. Crescenz VA Medical Center (CMCVAMC) is a national call center, study subjects (non-Veterans and Veterans) will be from all parts of the United States.

Family members (spouses, siblings, or parents) of Veteran will be recruited from Coaching Into Care, and offered telephone-based coaching to the family member regarding their concern that the Veteran has a substance abuse problem and does not want to seek treatment. The program will involve approximately 12 telephone calls over 4-6 months. Family members will be assessed for their own mental health symptoms, their perception of their Veteran's mental health symptoms and substance use, his or her treatment, as well as their perception of burden on the relationship with the Veteran. These assessments will occur at study entry, 6 months, and 12 months after study entry. Veteran's perceptions of the intervention will be sought at 12 months, whenever safe and practical. For Veterans who are not approached to participate in the study, VHA administrative data will be sought through a HIPAA Waiver to confirm any possible mental health and or substance abuse treatment the Veteran has received. Rates of initiation of treatment will be compared to QA data from the Coaching Into Care call center.

ELIGIBILITY:
Inclusion Criteria:

* CSO is a sibling, spouse/ intimate partner, or parent of a US military Veteran who served in Iraq or Afghanistan since 2001
* by the report of the CSO the Veteran of interest has a substance abuse problem that has led to interpersonal, legal, occupational, and/or health related negative consequences
* the CSO reports that the Veteran is not currently receiving treatment for this problem
* the CSO has contact 4+times/week and lives with or within 30 min. of the Veteran.

Exclusion Criteria:

* CSO has a SUD (Form 90, see Measures)
* the Veteran is currently incarcerated
* the CSO has no computer or other device with Internet access able to view video content
* the CSO or Veteran likely has a psychotic disorder (CSO report on the MINI) (see Measures)
* the CSO's involvement in a "coaching" intervention meant to encourage the Veteran to actively consider to seek care places the CSO at risk on a physical or psychological basis
* Callers who do not have access to a safe phone line will not be referred to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Sayers, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epidemiology Program: Post-Deployment Health Group, Analysis of VA Health Care Utilization among Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) Veterans: Cumulative from 1st Qtr FY 2002 through 4th Qtr FY 2014 (October 1, 2001 - September 30, 2014), Office of Public Health, Editor. 2015, Department of Veterans Affairs: Washington, DC. https://www.publichealth.va.gov/docs/epidemiology/healthcare-utilization-report-fy2015-qtr1.pdf
- [Background] Seal KH, Cohen G, Waldrop A, Cohen BE, Maguen S, Ren L. Substance use disorders in Iraq and Afghanistan veterans in VA healthcare, 2001-2010: Implications for screening, diagnosis and treatment. Drug Alcohol Depend. 2011 Jul 1;116(1-3):93-101. doi: 10.1016/j.drugalcdep.2010.11.027. Epub 2011 Jan 31. PMID 21277712
- [Background] Hearne CR. Predictors of Operation Enduring Freedom/Operation Iraqi Freedom veterans' engagement in mental health treatment. Mil Med. 2013 Nov;178(11):1183-7. doi: 10.7205/MILMED-D-13-00245. PMID 24183763
- [Background] Kim PY, Thomas JL, Wilk JE, Castro CA, Hoge CW. Stigma, barriers to care, and use of mental health services among active duty and National Guard soldiers after combat. Psychiatr Serv. 2010 Jun;61(6):582-8. doi: 10.1176/ps.2010.61.6.582. PMID 20513681
- [Background] Vogt D, Fox AB, Di Leone BA. Mental health beliefs and their relationship with treatment seeking among U.S. OEF/OIF veterans. J Trauma Stress. 2014 Jun;27(3):307-13. doi: 10.1002/jts.21919. Epub 2014 May 16. PMID 24839077
- [Background] Stinson FS, Grant BF, Dawson DA, Ruan WJ, Huang B, Saha T. Comorbidity between DSM-IV alcohol and specific drug use disorders in the United States: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Drug Alcohol Depend. 2005 Oct 1;80(1):105-16. doi: 10.1016/j.drugalcdep.2005.03.009. Epub 2005 Apr 18. PMID 16157233
- [Background] Batten S, Drapalski L, Decker L, DeViva C, Morris J, Mann A, Dixon B. Veteran interest in family involvement in PTSD treatment. Psychol Serv. 2009 Aug 10;6(3):184-189. doi: 10.1037/a0015392. PMID 30328689
- [Background] Hershenberg R, Mavandadi S, Klaus JR, Oslin DW, Sayers SL. Veteran preferences for romantic partner involvement in depression treatment. Gen Hosp Psychiatry. 2014 Nov-Dec;36(6):757-9. doi: 10.1016/j.genhosppsych.2014.08.001. Epub 2014 Aug 16. PMID 25219288
- [Background] Sayers SL, White T, Zubritsky C, Oslin DW. Family involvement in the care of healthy medical outpatients. Fam Pract. 2006 Jun;23(3):317-24. doi: 10.1093/fampra/cmi114. Epub 2006 Feb 3. PMID 16461451
- [Background] Marlowe DB, Merikle EP, Kirby KC, Festinger DS, McLellan AT. Multidimensional assessment of perceived treatment-entry pressures among substance abusers. Psychol Addict Behav. 2001 Jun;15(2):97-108. doi: 10.1037//0893-164x.15.2.97. PMID 11419236
- [Background] Sayers SL, Hess TH, Whitted P, Straits-Troster KA, Glynn SM. Coaching Into Care: Veterans Affairs Telephone-Based Service for Concerned Family Members of Military Veterans. Psychiatr Serv. 2021 Jan 1;72(1):107-109. doi: 10.1176/appi.ps.201900113. Epub 2020 Nov 10. PMID 33167815
- [Background] Meyers RJ, Roozen HG, Smith JE. The community reinforcement approach: an update of the evidence. Alcohol Res Health. 2011;33(4):380-8. PMID 23580022
- [Background] Roozen HG, de Waart R, van der Kroft P. Community reinforcement and family training: an effective option to engage treatment-resistant substance-abusing individuals in treatment. Addiction. 2010 Oct;105(10):1729-38. doi: 10.1111/j.1360-0443.2010.03016.x. PMID 20626372
- [Background] McKay JR, Van Horn D, Oslin DW, Ivey M, Drapkin ML, Coviello DM, Yu Q, Lynch KG. Extended telephone-based continuing care for alcohol dependence: 24-month outcomes and subgroup analyses. Addiction. 2011 Oct;106(10):1760-9. doi: 10.1111/j.1360-0443.2011.03483.x. Epub 2011 Aug 8. PMID 21545667
- [Background] McKay JR, Van Horn DH, Oslin DW, Lynch KG, Ivey M, Ward K, Drapkin ML, Becher JR, Coviello DM. A randomized trial of extended telephone-based continuing care for alcohol dependence: within-treatment substance use outcomes. J Consult Clin Psychol. 2010 Dec;78(6):912-23. doi: 10.1037/a0020700. PMID 20873894
- [Background] McKay JR, Lynch KG, Shepard DS, Ratichek S, Morrison R, Koppenhaver J, Pettinati HM. The effectiveness of telephone-based continuing care in the clinical management of alcohol and cocaine use disorders: 12-month outcomes. J Consult Clin Psychol. 2004 Dec;72(6):967-79. doi: 10.1037/0022-006X.72.6.967. PMID 15612844
- [Background] Erbes CR, Kuhn E, Polusny MA, Ruzek JI, Spoont M, Meis LA, Gifford E, Weingardt KR, Campbell EH, Oleson H, Taylor BC. A Pilot Trial of Online Training for Family Well-Being and Veteran Treatment Initiation for PTSD. Mil Med. 2020 Mar 2;185(3-4):401-408. doi: 10.1093/milmed/usz326. PMID 31621884
- [Background] Miller WR, Del Boca FK. Measurement of drinking behavior using the Form 90 family of instruments. J Stud Alcohol Suppl. 1994 Dec;12:112-8. doi: 10.15288/jsas.1994.s12.112. PMID 7722987
- [Background] Del Boca, F.K. and J.M. Brown, Issues in the development of reliable measures in addictions research: Introduction to Project MATCH assessment strategies. Psychology of Addictive Behaviors, 1996. 10(2): p. 67-74.
- [Background] Tonigan JS, Miller WR, Brown JM. The reliability of Form 90: an instrument for assessing alcohol treatment outcome. J Stud Alcohol. 1997 Jul;58(4):358-64. doi: 10.15288/jsa.1997.58.358. PMID 9203116
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Martin A, Rief W, Klaiberg A, Braehler E. Validity of the Brief Patient Health Questionnaire Mood Scale (PHQ-9) in the general population. Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):71-7. doi: 10.1016/j.genhosppsych.2005.07.003. PMID 16377369
- [Background] Oslin DW, Ross J, Sayers S, Murphy J, Kane V, Katz IR. Screening, assessment, and management of depression in VA primary care clinics. The Behavioral Health Laboratory. J Gen Intern Med. 2006 Jan;21(1):46-50. doi: 10.1111/j.1525-1497.2005.0267.x. PMID 16423122
- [Background] Oslin DW, Sayers S, Ross J, Kane V, Ten Have T, Conigliaro J, Cornelius J. Disease management for depression and at-risk drinking via telephone in an older population of veterans. Psychosom Med. 2003 Nov-Dec;65(6):931-7. doi: 10.1097/01.psy.0000097335.35776.fb. PMID 14645769
- [Background] Pinto-Meza A, Serrano-Blanco A, Penarrubia MT, Blanco E, Haro JM. Assessing depression in primary care with the PHQ-9: can it be carried out over the telephone? J Gen Intern Med. 2005 Aug;20(8):738-42. doi: 10.1111/j.1525-1497.2005.0144.x. PMID 16050884
- [Background] Savundranayagam MY, Montgomery RJ, Kosloski K. A dimensional analysis of caregiver burden among spouses and adult children. Gerontologist. 2011 Jun;51(3):321-31. doi: 10.1093/geront/gnq102. Epub 2010 Dec 6. PMID 21135026
- [Background] Weathers, F.W., J.A. Huska, and T.M. Keane, PCL-C for DSM-IV. 1991, Boston: National Center for PTSD - Behavioral Science Division.
- [Background] Rosner, B., Fundamentals of Biostatistics. 2011, Boston: Brooks/Cole.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited from the callers who reached a staff member of the Coaching Into Care (CIC) program. Those interested in considering the research study were screened by a study staff member, consented if eligible, and given a baseline assessment. Some participants responded to notices on social media who filled out a brief online screener or contact study staff directly. The matched TAU control participants were selected from callers to CIC in the same time period.
Groups:
- Coaching + VA-CRAFT: The interventionist provided a telephone-guided coaching intervention with the aid of a web-based program, VA-CRAFT, developed by the Co-Investigators for concerned significant others (CSOs). The VA-CRAFT program, based on the original Community Reinforcement and Family Training (CRAFT) program for substance misuse has 8 modules: 1) Introduction to CRAFT, 2) Overview of CRAFT, 3) Getting Started with CRAFT: Safety Planning, 4) Understanding substance abuse, 5) How to respond to substance abuse, 6) How to rebuild your life together, 7) How to help someone consider treatment, 8) Wrapping up. The goals of the intervention include helping the CSO understand triggers and long-term reinforcement of substance misuse, ignoring unhealthy behaviors and rewarding healthy behaviors, getting support, and encouraging the Veteran to enter mental health treatment for substance abuse. After viewing each of the VA-CRAFT web-based modules, the interventionist reviewed and personalized the material with the CSO via a telephone conversation. The intervention was flexible within the following framework: 1) 8 to 12, 30-45 min. telephone sessions, every 2-3 weeks, and 2) between 4 and 6 months.
- Treatment as Usual (TAU) Coaching: The treatment as usual coaching (TAU) seeks to empower, motivate, educate, and improved the concerned significant others' (CSOs') listening and communication skills with the goal of enhancing the veteran's intrinsic motivation for care. It draws from self-determination theory and emphasizes humans' underlying need for autonomy to maximize intrinsic motivation. CSOs were encouraged to reduce their pressure on the veteran to seek care and to engage in more positive activities of interest to both. CSOs were coached to listen for concerns expressed by the veteran, such as complaints about mood, anxiety, or the future (11, 12). CSOs were also encouraged to use an "autonomy-supportive" style of communication, which means offering to help the veteran but stating that it is understood that the offer is subject to the veteran welcoming this assistance. Coaching includes behavioral rehearsal to enhance the learning of these skills.
Period: Overall Study
Arm/Group | Coaching + VA-CRAFT | Treatment as Usual (TAU) Coaching
Started | 26 | 26
Completed | 15 (15 participants completed either 6-month or 12-month follow-up or both.) | 26 (Follow-up was limited to chart follow-up in CIC services)
Not Completed | 11 | 0
Not completed — deemed ineligible and administratively withdrawn | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coaching + VA-CRAFT | Treatment as Usual (TAU) Coaching | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: Age reported of caller participant (CSO) reported for Coaching + VA CRAFT group only. Age not assessed for TAU Coaching group (usual care).
  years
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 37.6 (7.9) |  | 37.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was not assessed for CSO's included in the TAU matched comparison group since race was not collected as part of usual clinical operations. Population: Race was not collected as part of TAU data collection for clinical purposes.
  Participants
    number analyzed (Participants) | 26 | 0 | 26
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 1 | 0 | 1
    White | 23 | 0 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Veteran's engagement in MH Care at Baseline [Count of Participants; unit: Participants] — As reported by CSO, the engagement of Veteran in MH Care at the baseline assessment, also reflecting that the Veteran was not engaged in MH care within the previous 6 months prior to the onset of study period.
  Participants | 0 | 0 | 0
Relationship [Count of Participants; unit: Participants] — Relationship of CSO to the Veteran: spouse/intimate other, sibling, parent
  Participants
    Spouses/intimate other | 21 | 20 | 41
    Sibling | 1 | 1 | 2
    Parent | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Veteran's Engaged in Mental Health Care
Description: Veteran's mental health care engagement was assessed from CSO participants' report.
Time Frame: At any point during study involvement, up to 1 year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Coaching + VA CRAFT | Treatment as Usual
Number analyzed (Participants) | 26 | 26
Participants | 7 | 5
Statistical Analysis 1: Comparison: Coaching + VA CRAFT vs Treatment as Usual; Test type: Superiority; p > .05, Z test of independent proportions; Z test of proportions = 0.66

ADVERSE EVENTS:
Time Frame: The investigators assessed for adverse events for the 1 year duration of participation for every participant in the study.
Arm/Group | Coaching + VA CRAFT | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
The limitations of the design include that this was a pilot study with a primary goal of examining the feasibility of the intervention rather than determine the efficacy of the intervention. The treatment as usual comparison group served only as a benchmark for understanding the potential effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT03246646/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03246646/ICF_001.pdf